CLINICAL TRIAL: NCT02161809
Title: Turn up the HEAT - Healthy Eating and Activity Time in Summer Day Camps
Acronym: HEPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Michael Beets, Principal Investigator, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00032881
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Childhood Obesity
Keywords: MVPA; Healthy Eating; children; childhood obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Diet, Healthy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Activity Intervention (Experimental): This arm (10 summer day camps) will receive the Physical Activity intervention the first year and both healthy eating and physical activity the second and thrid years.
  Interventions: Behavioral: Healthy Eating and Physical Activity
- Healthy EAting Intervention (Other): This arm (10 summer day camps) will receive the Healthy Eating intervention the first year and both healthy eating and physical activity the second and thrid years.
  Interventions: Behavioral: Healthy Eating and Physical Activity

INTERVENTIONS:
Behavioral: Healthy Eating and Physical Activity — The Healthy Eating and Physical Activity (HEPA) intervention aims to increase the quality of foods and beverages and physical activity opportunities in summer day camps. Through staff-level training, physical activity opportunities are modified to provide children with a substantial amount of meaningful physical activity. Through working with foods service providers, changes to the types of foods and beverages served will be made.
  Other Names: HEPA

SUMMARY:
The investigators long-term goal is to increase the number of Summer Day Camps (SDC) that meet the National Afterschool Association Healthy Eating and Physical Activity (HEPA) Standards. The objective is to evaluate the effectiveness of a multi-component intervention designed to increase children's PA levels and improve the quality of lunches and snacks children consume in SDCs. The HEPA intervention is designed to target children, parents, staff, program leaders, and the SDC environment and uses a train-the-trainer model with SDC leaders to train their staff to deliver and integrate the intervention into routine practice. In the proposed study, the investigators will evaluate these HEPA strategies, using a 4-year randomized controlled trial with 20 SDCs. An important feature of the study will be the evaluation of maintenance of the intervention after the removal of research support (e.g., training, boosters) during the final year, as well as costs associated with implementation.

The investigators hypothesize that intervention SDCs will achieve significantly greater increases in HEPA, compared to control SDCs. The investigators expect the study to support the cost-effectiveness and maintenance of our strategies for promoting HEPA that will facilitate SDCs meeting newly-established HEPA standards for this setting.

DETAILED DESCRIPTION:
The investigators aim to:

Evaluate the impact of the HEPA interventions on: 1.) The proportion of children meeting the PA Standard (i.e., ≥60min MVPA/d) while attending summer day camp; 2.) The proportion of foods (e.g., fruit, vegetable, water) children and staff bring and consume at the summer day camp that meet the HE Standards; and 3/) Changes in children's age-sex specific BMI percentile from the start to end of summer

Evaluate the cost-effectiveness of the HEPA intervention

Evaluate the maintenance of the HEPA intervention in summer day camps

ELIGIBILITY:
Inclusion Criteria:

* Summer Day camps will be eligible if:
* They operate for at least 10 weeks during the summer
* They do not have any primary focus such as sports, art, or tutoring (must be a general camp)
* Enrollment is at least 40 campers
* Operation hours are at least 8 hours.

Exclusion Criteria:

* Children will be unable to wear an activity monitor if experience any physical and/or orthopedic impairment that limits the child's ability to participate in regular PA (e.g., wheelchair user)

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2015-01; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Changes in percentage of children meeting 60min of MVPA | Year 1 - Year 4
  Changes in percentage of children at each summer day camp that meet the National Afterschool Alliance Standard of 60 minutes of moderate-to-vigorous physical activity daily.

SECONDARY OUTCOMES:
Change in percentage of children bringing/consuming healthy foods/beverages | Year 1 - Year 4
  Trained observers will record the foods/beverages brought/consumed at SDC - snacks and lunches

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Beets, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Weaver RG, Brazendale K, Chandler JL, Turner-McGrievy GM, Moore JB, Huberty JL, Ward DS, Beets MW. First year physical activity findings from turn up the HEAT (Healthy Eating and Activity Time) in summer day camps. PLoS One. 2017 Mar 28;12(3):e0173791. doi: 10.1371/journal.pone.0173791. eCollection 2017. PMID 28350830